CLINICAL TRIAL: NCT02463487
Title: Negative Pressure Wound Therapy as a Drug Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Larry Lavery, Professor, Department of Plastic Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 092014-016
Record Dates: First submitted 2015-04-16; First posted 2015-06-04 (Estimated); Results first posted 2020-08-14 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Negative-Pressure Wound Therapy; Therapeutic Irrigation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cardinal Pro + Irrigation (NPWTi) (Active Comparator): Negative Pressure Wound Therapy with Irrigation: Quantum™ +Simultaneous Irrigation (NPWTi) - Negative Pressure Wound Therapy with Prontosan® Intervention is receiving the Cardinal Vac with Irrigation
  Interventions: Device: Cardinal Pro +Simultaneous Irrigation (NPWTi)
- Cardinal Pro (NPWT) Therapy (Active Comparator): Negative Pressure Wound Therapy without Irrigation: Quantum™ (NPWT) -Negative Pressure Wound Therapy (without Prontosan®) Intervention is receiving the Cardinal Vac without Irrigation
  Interventions: Device: Cardinal Pro (NPWT) Therapy

INTERVENTIONS:
Device: Cardinal Pro +Simultaneous Irrigation (NPWTi) — NPWT with low volume irrigation (15 cc/hr) with 1% polyhexanide biguanide (PHMB), Prontosan®
  Other Names: • Negative Pressure Wound Therapy with Irrigation
  Arms: Cardinal Pro + Irrigation (NPWTi)
Device: Cardinal Pro (NPWT) Therapy — NPWT 125 mm Hg continuous pressure with foam interface
  Other Names: • Negative Pressure Wound Therapy without Irrigation
  Arms: Cardinal Pro (NPWT) Therapy

SUMMARY:
The investigators plan a randomized clinical trial of 150 patients with infected diabetes-related lower extremity wounds to compare the clinical and economic effectiveness of negative pressure wound therapy with continuous irrigation and negative pressure wound therapy without irrigation.

DETAILED DESCRIPTION:
The investigators will enroll 150 patients from two centers: The University of Texas Southwestern University Hospital and Parkland Hospital. The investigators will screen and enroll patients with wounds in the inpatient setting. Patients will be randomized to receive traditional NPWT or NPWT with continuous irrigation while they are hospitalized. The average hospitalization for patients that receive NPWT is 13.3 days. Patients that do not have their wound surgically closed during hospitalization will be discharged with negative pressure wound therapy for up to a total of four weeks of therapy. After discharge from the hospital, subjects will be seen twice weekly by home health, and will be evaluated in clinic every 7 days (±7 days) up to a total of 16-week period or until 30 days after the wound heals.

Study Procedures:

Screening Procedures

* Review and sign the Informed Consent and HIPAA Authorization
* The study doctor will review the inclusion and exclusion criteria
* Demographics (such as age, gender, race or ethnicity)
* Physical exam
* Sitting blood pressure and pulse
* Height and weight
* Collection of the medical and surgical history
* Collection of the history of the wound
* Wound assessment(s)/Debridement - various tests and measurements to assess the sensation (feeling) and circulation (blood flow) in the subject's feet and lower legs. None of these tests are invasive (using needles), uncomfortable or have risks greater than standard care.
* Wound imaging - photographs and images of the subject's wound using acetate tracings, a digital camera and an ARANZ camera (a special type of camera that uses computer software to calculate the volume of the wound)
* Hyperspectral imaging
* Vascular/Neurological evaluation
* Results of standard-of-care laboratory tests including a white blood cell count, blood chemistry (tests to see how well organs, such as the liver and kidneys are working), and blood glucose. Results of a serum pregnancy test (standard care for women of child-bearing potential as part of pre-op labs) will also be collected. About 2 tablespoons of blood will be drawn for these tests.
* Collection of a list of the subject's current medications, including prescriptions, over-the-counter medications, supplements and herbals.

This visit will last about 2 hours.

If the subject qualifies for the study, they will participate in the following procedures:

Group Assignment

If the researchers believe the subject can take part in this study, s/he will be assigned randomly (like a flip of a coin) to receive one of the following therapies:

* Negative Pressure Wound Therapy with Irrigation
* Negative Pressure Wound Therapy without Irrigation

The group is assigned randomly (like flipping a coin). The sponsor or researchers do not know in advance what group assignment each subject will receive. Neither the subject nor the researchers will be allowed to choose which group s/he is assigned to.

Study Intervention

The subject will receive either:

* Cardinal Pro +Simultaneous Irrigation (NPWTi) - Negative Pressure Wound Therapy with Prontosan®, or
* Cardinal Pro (NPWT) Therapy (without Prontosan®)

Assigned therapy will continue in the hospital until the physician determines that the wound is ready for closure. If the subject's wound is healing, study therapy will be discontinued and standard dressings will be applied. If surgical closure is needed, the subject will return to the Operating Room for a procedure to close the wound.

If the wound is not ready for closure during the hospital stay, subjects will continue NPWT at home for the remainder of the 4 weeks of treatment. NPWT at home will be without irrigation (KCI VAC Via®).

Procedures and Evaluations during the Research The study therapy will only be given while the subject is in the hospital. S/he will continue the therapy for up to 4 weeks or until the wound is closed. Once the therapy is stopped s/he will continue to be followed by the study doctor. After the subject is released from the hospital s/he will need to see the study doctor Every 7 days (±7 days). If the subject's wound does not heal before 56 days after his/her first surgery then s/he will no longer be taking part in the study. The study doctor will continue to check the wound. If the wound closes, s/he will see the study doctor 30 days later to have the closed wound checked.

12 Month Extension:

After the end of the defined study period, the patients will be followed observationally by their electronic medical records for 12 months as it would not be feasible to ask them to return for an in-person evaluation as: patients have moved, no longer have correct contact information, as well as it would create a financial hardship on the patients to return for further visits. In order to more appropriately determine long term results from participation, a longer period of time of follow up is necessary. Related outcomes that we would like to follow over a 12-month duration are incidence of new foot ulcerations, re-ulceration of a previously healed foot wound, healing and time to healing of patients who took longer than the current study allows, duration of antibiotics received for foot infections, re-admissions to the hospital, need for subsequent surgery, amputation, loss of limb, and death. This expanded follow up period would provide valuable information to the long-term outcomes and complications of this high risk population and will help direct how future efforts may be better focused to reduce complications and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of diabetes mellitus Men/women ≥21 years old Foot or ankle wounds sized 5 cm2 -100 cm2 ABI≥0.5 or toe pressures >30 mmHg

Exclusion Criteria:

Active Charcot arthropathy Unable to use NPWT at home Untreated bone or soft tissue infection Unable to keep research appointments Active alcohol or substance abuse

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Lavery LA, Davis KE, La Fontaine J, Farrar JD, Bhavan K, Oz OK, Crisologo PA. Does negative pressure wound therapy with irrigation improve clinical outcomes? A randomized clinical trial in patients with diabetic foot infections. Am J Surg. 2020 Oct;220(4):1076-1082. doi: 10.1016/j.amjsurg.2020.02.044. Epub 2020 Feb 27. PMID 32139102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was comprised of patients who were admitted to hospital with a moderate or severe foot infection that required incision and drainage and parenteral antibiotics and for whom negative pressure wound therapy (NPWT) was indicated. Patients who fit the criteria for the study were then recruited.
Pre-assignment Details: The patients underwent a screening exam including
  * evaluating sensory neuropathy with loss of protective sensation with a 10-gram monofilament
  * Vibration Perception Threshold Testing
  * ABI - ankle brachial index
  * SPP - skin perfusion pressure
  * Peripheral arterial disease (PAD) was defined as either ABI <0.9 or SPP <30 mm Hg.
Period: Overall Study
Arm/Group | Cardinal Pro + Irrigation (NPWTi) | Cardinal Pro (NPWT) Therapy
Started | 75 | 75
Completed | 65 | 65
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardinal Pro (NPWT) Therapy | Cardinal Pro + Irrigation (NPWTi) | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.32 (8.22) | 49.07 (9.74) | 50.19 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 58 | 59 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 21 | 18 | 39
  Native American | 1 | 1 | 2
  African American | 30 | 30 | 60
  Hispanic | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Complete Healing or Coverage of the Study Wound
Description: How many wounds fully healed in 16 weeks. Healing defined as fully epithelialized skin with no drainage.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cardinal Pro (NPWT) Therapy | Cardinal Pro + Irrigation (NPWTi)
Number analyzed (Participants) | 75 | 75
Participants | 44 | 45
Statistical Analysis 1: Comparison: Cardinal Pro (NPWT) Therapy vs Cardinal Pro + Irrigation (NPWTi); Test type: Other; p = 0.87, t-test, 1 sided

2. Secondary Outcome: Total Adverse Events of Participants
Description: Total number of adverse events, including new foot ulcer formation, all-cause hospital readmission, and foot-related hospital readmission.
Time Frame: 16 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cardinal Pro (NPWT) Therapy | Cardinal Pro + Irrigation (NPWTi)
Number analyzed (Participants) | 75 | 75
Participants
  New ulcer formation | 12 | 18
  All-cause readmission | 26 | 27
  Foot-related readmission | 13 | 14

3. Secondary Outcome: Number of Participants With Wound Dehiscence After Hospital Discharge
Description: Dehiscence is defined as any part of a surgically closed wound that failed to heal when sutures were removed.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cardinal Pro (NPWT) Therapy | Cardinal Pro + Irrigation (NPWTi)
Number analyzed (Participants) | 75 | 75
Participants | 46 | 40
Statistical Analysis 1: Comparison: Cardinal Pro (NPWT) Therapy vs Cardinal Pro + Irrigation (NPWTi); Test type: Other; p = 0.08, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Cardinal Pro (NPWT) Therapy | Cardinal Pro + Irrigation (NPWTi)
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 39/75 | 41/75
Other Adverse Events (participants affected / at risk) | 27/75 | 35/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cardinal Pro (NPWT) Therapy (N=75) | Cardinal Pro + Irrigation (NPWTi) (N=75)
All-cause hospital readmission (Surgical and medical procedures) | 26 | 27 — Readmission to hospital for any reason after initial discharge
Foot-related hospital readmission (Infections and infestations) | 13 | 14 — Readmission to the hospital after initial discharge for foot related infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cardinal Pro (NPWT) Therapy (N=75) | Cardinal Pro + Irrigation (NPWTi) (N=75)
New ulcer formation (Skin and subcutaneous tissue disorders) | 12 | 18 — Formation of foot ulcer (different than the index ulcer) during the study
Reinfection (Infections and infestations) | 15 | 17 — Reinfection of the ulcer on the study foot

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02463487/Prot_SAP_000.pdf